CLINICAL TRIAL: NCT03061383
Title: Reduction of Dentine Hypersensitivity Using 8% Arginine Based Toothpaste and 8% Strontium Acetate Based Toothpaste: Randomized Controlled Clinical Trial
Brief Title: Reduction of Dentine Hypersensitivity Using 8% Arginine Based Toothpaste and 8% Strontium Acetate Based Toothpaste (DH)
Acronym: DH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Abdel Ghaffar Ahmed Ali, Reduction of dentine hypersensitivity using 8% Arginine based toothpaste and 8% Strontium acetate based toothpaste: Randomized Controlled clinical trial, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEBC-CU-2017-02-16
Record Dates: First submitted 2017-02-19; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Dentin Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Intervention Model Description: Participants will be tested in this study having at least 3 sensitive sound teeth. Participants will be divided into 3 groups, according to the type of desensitizing agents (D); D1 treatment using 8% arginine based toothpaste (Colgate Pro-relief), D2 treatment using 8% strontium acetate based toothpaste (Sensodyne Rapid Action) and D3 control group using placebo (gel without any active ingredient).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: It will be a triple blinded study so that the participant, the researcher and the data analysis will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 8% Arginine based toothpaste (Active Comparator): The procedure will be performed after scaling in group D1 using 8% arginine based toothpaste (Colgate Pro-relief) . Treatment will be done at baseline then patients will use the toothpaste at home twice per day by using soft bristled tooth brush and the given dentifrice using modified stillmans method as explained by examiner
  Interventions: Other: 8% Arginine based toothpaste
- 8% Strontium acetate based toothpaste (Active Comparator): The procedure will be performed after scaling in group D2 using 8% strontium acetate based toothpaste (Sensodyne Rapid Action) . Treatment will be done at baseline then patients will use the toothpaste at home twice per day by using soft bristled tooth brush and the given dentifrice using modified stillmans method as explained by examiner
  Interventions: Other: 8% strontium acetate based toothpaste
- tooth past without active ingredient (Placebo Comparator): The procedure will be performed after scaling in group D3 control group using placebo . Treatment will be done at baseline then patients will use the toothpaste at home twice per day by using soft bristled tooth brush and the given dentifrice using modified stillmans method as explained by examiner
  Interventions: Other: placebo

INTERVENTIONS:
Other: 8% Arginine based toothpaste — toothpaste
  Other Names: Colgate sensitive Pro-relief
  Arms: 8% Arginine based toothpaste
Other: 8% strontium acetate based toothpaste — toothpaste
  Other Names: Sensodyne Rapid Action
  Arms: 8% Strontium acetate based toothpaste
Other: placebo — toothpaste
  Arms: tooth past without active ingredient

SUMMARY:
This is a randomized, triple-blind, placebo-controlled study. 51 subjects with a confirmed diagnosis of dentin hypersensitivity were randomized to one of three treatments: Arginine based toothpaste, strontium acetate based toothpaste , or placebo. Treatment will be done at baseline then patients will use the toothpaste at home twice per day by using soft bristled tooth brush and the given dentifrice using modified stillmans method as explained by examiner. Standard test stimuli is calibrated short blast of air syringe, will be applied to sensitive dentin surfaces. Subjects recorded the intensity of sensitivity in response to stimulus on a visual analog scale at baseline, and after 1 week, 2 weeks and 3 months.

DETAILED DESCRIPTION:
* Study setting This study will be carried out on adult patients attending to the operative clinic in The Faculty of Oral and Dental Medicine, Cairo University, Egypt. The procedures will be carried out by postgraduate student esraa abdel ghaffar ahmed ali [B.D.S. 2012 from Misr International University] without an assistant.
* Eligibility criteria

  * Inclusion criteria Normal adults will be recruited in this study, all the volunteers participated in this experiment will be healthy looking with free medical history.

Subjects aged between 18-35 years At least three sensitive teeth (buccal /facial) aspect with recession , abrasion, erosion with a score of >3 on verbal rating scale, ranging from 0-3= no pain/mild pain, 4-6= moderate pain, and 7- 10= severe pain. Subjects were required to be available for the duration of the study, and to sign an informed consent form

-Exclusion criteria Subjects with a history of allergy to any of the drugs or chemicals used in the study.

Any removable appliance (RPD or orthodontic retainer). Ongoing orthodontic treatment with fixed appliances.

Presence of any large or defective restorations, cracked enamel or caries on the hypersensitive tooth.

Pregnancy and lactating mothers. Dental pathology causing pain similar to dentin hypersensitivity. Patients with any systemic problem or mental or physical disability

-Grouping of participants: Participants will be tested in this study having at least 3 sensitive sound teeth. Participants will be divided into 3 groups, according to the type of desensitizing agents (D); D1 treatment using 8% arginine based toothpaste (Colgate Pro-relief), D2 treatment using 8% strontium acetate based toothpaste (Sensodyne Rapid Action) and D3 control group using placebo (gel without any active ingredient).

-Intervention : The procedure will be performed after scaling in group D1 using 8% arginine based toothpaste (Colgate Pro-relief) , group D2 using 8% strontium acetate based toothpaste (Sensodyne Rapid Action) and D3 control group using placebo . Treatment will be done at baseline then patients will use the toothpaste at home twice per day by using soft bristled tooth brush and the given dentifrice using modified stillmans method as explained by examiner. The choice of the following brushing method was made on its well established efficiency to clean the sulcular areas which is a potential niche for plaque accumulation. Dental plaque is itself considered as one of the possible cause of dentin hypersensitivity. Additionally Modified Stillmans technique is shown to increase the gingival crevice fluid flow thus providing a flushing action. Patient will be recalled after 1 week , 2 weeks and 3 months for evaluation the effect of intervention on reduction of dentin hypersensitivity . The application procedures will follow manufacturer's instructions.

-Testing procedures: Dentinal hypersensitivity will be measured using a Visual Analogue Scale (VAS) to record the response from a calibrated short blast of air syringe at the four time intervals "baseline, 1 week , 2 weeks and 3 months"

-Randomization: Randomization will be done according to a check list done by a dentist other than the researcher including the number of participants divided into 3 subgroups denoting with letter A, B and C.

-Sample size calculation: This study will be conducted to evaluate the effect of 8% arginine based toothpaste in comparison to 8% strontium acetate based toothpaste on dentin hypersensitivity reduction. Based on the previous study by SHAH 2015, the mean dentine hypersensitivity was 3.3+_ 0.6 in Colgate paste and 2.6 +_ 0.7 for Sensodyne past. Using power 80% and 5% significance level, 15 patients in each group will be sufficient. This number is to be increased to 17 patients to compensate for possible losses during follow up. The sample size was calculated by G power.

-Recruitment Announcement to residents of outpatient clinic in Conservative Dentistry- Faculty of Oral and Dental Medicine- Cairo University Egypt, to screen adult patient during diagnosis for their chief complain so patients with at least three sensitive teeth will be enrolled in this study, if they meet the eligibility criteria.

-Allocation

1. sequence generation Randomization is done by computer software www.random.org. The sequence generates 3 codes (A, B and C).
2. Allocation and concealment arrangement A checklist will be designed by a dentist other than the researcher to identify each material specimen
3. Implementation Allocation sequence will be generated at the Center of Evidence Based Dentistry, Faculty of Oral and Dental Medicine - Cairo University.

   Participant enrollment will be done by the principle investigator
   * Blinding:

   It will be a triple blinded study so that the participant, the researcher and the data analysis will be blinded.
   * Data collection methods:

   There will be a file for each participant includes his/her( informed consent, the 4 time interval visual analogue scale, all data including address, phone numbers) and all information that will be needed for follow up.
   * Retention In order to ensure that the participants will come back for the sequence visits, the patient will be asked for the telephone number and address and will be called before the visit.

   Explanation of the importance of the study is explained to patient and the importance on keeping the appointments

   -Data management Explain to the patient the importance of this study and that commitment to the appointments is mandatory to get the best results from this study.

   All data is documented in the patient sheet. -Statistical Methods Data will be analyzed using IBM SPSS advanced statistics (Statistical Package for Social Sciences), version 21 (SPSS Inc., Chicago, IL). Numerical data will be described as mean and standard deviation or median and range. Data will be explored for normality using kolmogorov - Smirnov test and Shapiro-Wilk test. Comparisons between 3 groups for normally distributed numeric variables will be done using the ANOVA while for non normally distributed numeric variables will be done by Kruskal Wallis test. A p-value less than or equal to 0.05 will be considered statistically significant. All tests will be two tailed.

   Categorical data will be described as numbers and percentages and comparisons will be done by chi square test or fisher exact as appropriate.

   -Data Monitoring This study will be monitored by the supervisors who will have full access to the results and will take the final decision to terminate the trial.

   -Harms No reported adverse effect of both interventions was reported. In case of any harm during the trial it will be reported, documented and treated.

   -Auditing Auditing of the study design will be done by the evidence based committee- Faculty of Oral and Dental Medicine- Cairo University.

   -Ethics and dissemination Patient consent. Detailed check list including the exact procedure and interventions that will be performed, the number of visits, the importance of this study to the participants, as well as its importance to the population, and the possible adverse effects accompanied with the use of the intervention.

   -Research ethics approval This protocol and the template of informed consent form will be reviewed by the Ethics Committee of scientific research, Faculty of Oral and Dental Medicine- Cairo University.

   -Protocol amendments Any modifications to the protocol which may have an impact on the conduction of the study, potential benefit of the patient or may affect the patient safety, including changes of study objectives, study design, sample size, study procedure or significant administrative aspects will require a formal amendment to the protocol. Such amendment will be agreed upon by the council of Conservative dentistry Department.

   -Consent and assent Researcher will discuss the trial with the participant's. They will be able to discuss his thoughts with the researcher after a full explanation of the procedure in simple words. A verbal assent will be taken from the participating patient while a written consent is signed by the patient.

   -Confidentiality All study related information will be stored securely. All participants'' information will be stored in a locked file cabinets in areas with limited access. Process and administrative forms will be identified by a coded ID [identifier number] only to maintain participants' confidentiality. All records that contain names or other personal identifiers will be stored separately from study records identified by code number.

   -Declaration of interest Non-financial
   * Access to data All principle investigators will be given access to the data sets. All data sets will be password protected.
   * Ancillary and post-trial care Full mouth treatment will be offered to all the participants in addition to post-operative care and preventive measures after the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Normal adults will be recruited in this study, all the volunteers participated in this experiment will be healthy looking with free medical history.
* Subjects aged between 18-35 years
* At least three sensitive teeth (buccal /facial) aspect with recession , abrasion, erosion with a score of >3 on verbal rating scale, ranging from 0-3= no pain/mild pain, 4-6= moderate pain, and 7- 10= severe pain.
* Subjects were required to be available for the duration of the study, and to sign an informed consent form

Exclusion Criteria:

* Subjects with a history of allergy to any of the drugs or chemicals used in the study.
* Any removable appliance (RPD or orthodontic retainer). Ongoing orthodontic treatment with fixed appliances.
* Presence of any large or defective restorations, cracked enamel or caries on the hypersensitive tooth.
* Pregnancy and lactating mothers.
* Dental pathology causing pain similar to dentin hypersensitivity.
* Patients with any systemic problem or mental or physical disability

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2017-03-03 (Estimated); Primary Completion 2018-10-03 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
reduction of dentin hypersensitivity | 3 months
  Subjects recorded the intensity of sensitivity in response to stimulus on a visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: mohamed adel ezzat khairy, PHD, Study Director — Professor of Conservative Dentistry, Faculty of Oral and Dental Medicine, Cairo University; Maha abdel salam El-baz, PHD, Study Chair — Lecturer of Conservative Dentistry, Faculty of Oral and Dental Medicine, Cairo University
Locations (1):
- Esraa Abdel Ghaffar Ahmed Ali, Madīnat an Naşr, Egypt

IPD SHARING:
Plan to Share IPD: Yes
publishing the data at egyptian dental journal

REFERENCES:
- [Background] Pinto SC, Bandeca MC, Pinheiro MC, Cavassim R, Tonetto MR, Borges AH, Sampaio JE. Preventive effect of a high fluoride toothpaste and arginine-carbonate toothpaste on dentinal tubules exposure followed by acid challenge: a dentine permeability evaluation. BMC Res Notes. 2014 Jun 24;7:385. doi: 10.1186/1756-0500-7-385. PMID 24958423